CLINICAL TRIAL: NCT03587909
Title: Intraoperative Performance and Postoperative Outcomes Following Femtosecond Laser Assisted Cataract Surgery (FLACS) and Manual Phacoemulsification in Eyes With Shallow Anterior Chamber
Brief Title: FLACS vs Phaco in Shallow Anterior Chamber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Principal Investigator, Abhay R. Vasavada, Principal Investigator, Iladevi Cataract and IOL Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FLACS1
Record Dates: First submitted 2018-06-11; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Cataract Surgery; Shallow Anterior Chamber; Phacoemulsification
Keywords: FLACS; Phaco; Shallow Anterior Chamber

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phacoemulsification Cataract Surgery (Active Comparator): Procedure / Surgery : Phacoemulsification Surgery
  Interventions: Procedure: Phacoemulsification Cataract SUrgery
- Femtosecond Cataract Surgery (Active Comparator): Procedure / SUrgery - Femtosecond Laser Cataract surgery
  Interventions: Procedure: Femtosecond Cataract Surgery

INTERVENTIONS:
Procedure: Phacoemulsification Cataract SUrgery — Phacoemulsification in eyes with shallow anterior chamber (<2.5mm depth)
  Arms: Phacoemulsification Cataract Surgery
Procedure: Femtosecond Cataract Surgery — Femtosecond Cataract Surgery in eyes with shallow anterior chamber < 2.5mm
  Arms: Femtosecond Cataract Surgery

SUMMARY:
Phacoemulsification in eyes with a shallow anterior chamber (ACD < 2.2mm) presents with problems of safe access to the cataract and increased vulnerability of the endothelium and a higher tendency of complications such as descemet's detachment and iris prolapse. A shallow anterior chamber is also responsible for the high incidence of glaucoma and postoperative complications after cataract surgery. Femtosecond assisted cataract surgery has made cataract surgery safer and more predictable. The effective phacoemulsification time and intra-operative manipulation is greatly reduced in FLACS. However phacoemulsification still remains the most widely performed cataract surgery around the world. Post-operative outcomes after phacoemulsification in patients having shallow anterior chamber have been extensively reported in literature over the years.

There is no head to head comparison in terms of intraoperative performance and post-operative outcomes between FLACS and phacoemulsification in eyes with shallow anterior chamber.

The aim is to compare the intra-operative performance and post-operative outcomes in eyes undergoing femtosecond laser assisted cataract surgery versus eyes undergoing phacoemulsification in eyes having shallow anterior chamber.

The study will bring an understanding on the question: Do patients undergoing Femtosecond laser assisted cataract surgery behave differently from those undergoing phacoemulsification?

DETAILED DESCRIPTION:
Inclusion Criteria:

* Age-related cataract
* Shallow Anterior Chamber (<2.5mm)

Exclusion Criteria:

-Ocular co-morbidity - corneal disorders, glaucoma, uveitis, previous ocular surgery

Surgical Technique :

* Standardized, Single Surgeon
* 2.2 mm clear corneal temporal incision
* FLACS Group : Capsulorhexis, Lens Fragmentation with femto laser

The investigators will be evaluating the following parameters:

1. Primary outcome measure Corneal thickness on day 1, week 1 and 1 month (Change in corneal thickness of 15% from preop. will be considered significant).
2. Secondary outcome measures

   * Corneal clarity -on day 1, week 1 and 1 month postoperatively
   * Anterior chamber cells and flare (Hogan's criteria)
   * Percentage change in endothelial cell density from preoperatively to 3 months postoperatively
   * Unaided visual acuity (distance) on day 1 and 1 month.
   * Best corrected distance visual acuity 1 month postoperatively
3. Other Observations :

1) Cumulative Dissipated Energy (CDE) 2) Surgical time 3) Fluid used 4) Descemets membrane detachment during surgery 5) Incidence of iris trauma 6) Any other intra-operative complications

ELIGIBILITY:
Inclusion Criteria:

* uncomplicated, age related cataracts
* Shallow anterior chamber (measured as </=2.5mm )

Exclusion Criteria:

* Coexisting ocular morbidity,
* inability to come for followup

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Central Corneal Thickness | Postoperative Day 1
  Central Corneal Thickness

SECONDARY OUTCOMES:
Anterior Chamber Inflammation | Postoperative Day 1
  Anterior chamber cells and flare (Hogan's criteria)
Endothelial Cell Morphology | Postoperative 6 months
  Endothelial Cell Density

CONTACTS AND LOCATIONS:
Overall Officials: Abhay Vasavada, MS,FRCS, Principal Investigator — Iladevi Cataract & IOL Research Centre, Ahmedabad
Locations (1):
- Iladevi Cataract & IOL Research Center, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No